CLINICAL TRIAL: NCT07263893
Title: Evaluation of the Efficacy of Custom-Made Inter-flex Three-Dimensional Plate in Treatment of Mandibular Fracture A Randomized Controlled Clinical Trial
Brief Title: Inter Flex Three Dimensional Plate in Management of Mandibular Fracture RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/1012
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Mandibular Fracture Treatment
Keywords: INTER-FLEX 3D PLATE; mandibular fractures; radiographic assesment; time of surgery; healing
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: Brand name thickness Composition Company software Customized CAD CAM milled plates 1mm Titanium plate Arab engineers corporation blender Screws 2mm Titanium screw Arab engineers corporation blender
  II- Methods:
  1. Study Design: Randomized clinical study via www.randomizer.org
  2. Study Setting: This study will be conducted on twenty mandibular fracture sites
  3. Study population and sampling:
  Patients will be selected from the outpatient clinic of the Oral and Maxillofacial Surgery department in the Faculty of Dentistry, Suez Canal University also from emergency room of Mataria Teaching Hospital.
  All patients will be informed with all the details of the surgical procedures, complications and the whole study schedule. Then, each patient will sign an informed consent. Patients participating in the current study will have to fulfill the following eligibility criteria:
  Inclusion criteria: (Zhao et al., 2018)
  1-Patients who are suffering from re
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I: site with mandibular fracture will be treated with custom made Inter-flex three dimensional (Experimental): site with mandibular fracture will be reduced and fixation will be done .visibility using custom made Inter-flex three dimensional plate plates in Group I and fixation using custom made Inter-flex three dimensional according to champ's lines of osteo-synthesis in Group I. closure of the surgical field with vicryl suture material (90% glycolide and 10% L-lactide: Ethicon part of Johnson & Johnson Int, US.).
  Interventions: Procedure: Group I :site with mandibular fracture will be treated with custom made Inter-flex three dimensional plate in site of mandibular fracture
- Group II: site with mandibular fracture will be treated with a ready-made Titanium plates in site of (No Intervention): site with mandibular fracture will be reduced and fixation will be done .visibility using conventional double-mini plates in Group II and fixation using 2 mini-plates according to champ's lines of osteo-synthesis in Group II.

INTERVENTIONS:
Procedure: Group I :site with mandibular fracture will be treated with custom made Inter-flex three dimensional plate in site of mandibular fracture — site with mandibular fracture will be reduced and fixation will be done .visibility using custom made Inter-flex three dimensional plate plates in Group I and fixation using custom made Inter-flex three dimensional according to champ's lines of osteo-synthesis in Group I. closure of the surgical field with vicryl suture material (90% glycolide and 10% L-lactide: Ethicon part of Johnson & Johnson Int, US.).
  Arms: Group I: site with mandibular fracture will be treated with custom made Inter-flex three dimensional

SUMMARY:
The goal of this clinical trial is to learn if The use of a 3D-designed Inter-flex plate will achieve safe and desirable anatomical & functional restoration with reduced operative time in mandibular fracture,

* Improvement of occlusal and inter-cuspal relation in addition to stabilized intra-fragmentary mobility,
* Offer greatest resistance to displacement
* shows most favorable biomechanical behavior

DETAILED DESCRIPTION:
Mandibular fractures most commonly accompany facial trauma, with nearly half of the patients requiring surgical repair. The treatment of fractures prioritizes the restoration of functionality through The realignment of fractured segments. Conventional methods, such as titanium plates, have been employed for this purpose; however, certain limitations have been observed, such as there is a chance of potential infection and mal-union in mandibular fracture site. Leading to the development of patient specific plates. Furthermore, recent advancements in digital technology in Dentistry enable creation of virtual models and simulations of surgical Procedures. Aim: Is to evaluate the effect of custom-made Inter-flex three dimensional plate vs conventional ready-made Titanium plates in Management of Mandibular Fracture Methodology: This study will be conducted on 20 sites with mandibular fracture in patients. The sites of fracture will be divided into two groups (Group I and Group II) randomly and equally via www.randomizer.org Group I: site with mandibular fracture will be treated with custom made Inter-flex three dimensional plate in site of mandibular fracture, Group II: site with mandibular fracture will be treated with a ready-made Titanium plates in site of mandibular fracture. The postoperative clinical evaluation included presence of infection, stability of the mandibular lower border, state of occlusion, maximal mouth opening. Postoperative radiographic examinations to evaluate the accuracy of reduction and bony union using postoperative c.t 24hour and 3 months by measuring the inter-fragmentary gap and the Intergonial distance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are suffering from recent, uninfected, and minimally displaced or unfavorable mandibular fractures
2. Adult patients with no gender predilection that agreed to present for follow-up visits for minimum postoperative period of immediate,3 months,6 months.
3. A fracture that demands open reduction and internal fixation
4. Patients under ASA-1 category

Exclusion Criteria:

1. Comminuted, infected mandibular fracture.
2. Pediatric patients below 4 years old and geriatric patients with completely edentulous mouth.
3. Patient with osteoporosis
4. Medical compromised patient (Poorly controlled DM or HTN, COPD, morbid obesity (BMI ≥40), Recent (<3 months) MI, ongoing cardiac ischemia or severe valve dysfunction, severe reduction of ejection fraction, shock, sepsis, undergoing regularly scheduled dialysis, history (>3 months)
5. Fractures in completely edentulous patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation | 24 hour after surgery and after 3 months
  * The linear inter-fragmentary gap between the fractured segments in mm
  * Intergonial distance was measured between the most inferior, lateral, and posterior points of the mandible bilaterally as determined on CT in mm.
Mobility of fracture segments | 24 hour after surgery
  assessed through bimanual digital manipulation
  * Stable >> no movement of fragments.
  * Nonstable >> presence of movement.
State of occlusion | after 24 hours and after 3 months of surgery
  will be assessed by asking the patient to bite in maximum intercuspation at each follow-up (intact/deranged) also by recording molar relation as (satisfactory or deranged).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ah Elsholukamy, Professor, Study Director — Suez Canal University; Mohamed Na Gad Elhaq, lecturer, Study Director — Suez Canal University; Maurice Fe khalil, consultant, Study Director — Mataria Teaching Hospital
Locations (1):
- Mataria Teaching Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
because these are patient data that cant be shared

REFERENCES:
- [Result] Saad, A., Khalil, A. F., & El-Mahallawy, Y. (2025). INTERFLEX PLATE VERSUS CONVENTIONAL MINIPLATES IN THE MANAGEMENT OF ANTERIOR MANDIBULAR FRACTURES. a RANDOMIZED CONTROLLED CLINICAL TRIAL. Alexandria Dental Journal, 0(0), 0. https://doi.org/10.21608/adjalexu.2025.344361.1572
- See also: INTERFLEX PLATE VERSUS CONVENTIONAL MINIPLATES IN THE MANAGEMENT OF ANTERIOR MANDIBULAR FRACTURES. A RANDOMIZED CONTROLLED CLINICAL TRIAL — https://journals.ekb.eg/article_445927.html